CLINICAL TRIAL: NCT04556643
Title: Effectiveness of Breathing Exercises During the Second Stage of Labor on Labor Pain and Duration
Brief Title: Effectiveness of Breathing Exercises During the Second Stage of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00239 Maryam Waheed
Record Dates: First submitted 2020-09-16; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Labor Pain
Keywords: labor pain; Breathing Exercises; second stage of labor
MeSH Terms: conditions — Labor Pain | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Two sessions will be given to pregnant women in Intervention group. One session breathing exercises training will be given during first stage of labor by the investigator. During training all participants in Intervention group will be instructed to perform breathing exercises during the second stage of labor.
  Interventions: Other: Breathing exercises
- Control Group (No Intervention): Usual hospital delivery protocol will be followed.

INTERVENTIONS:
Other: Breathing exercises — The main components of breathing exercises during training will be as follows (A) First, fill your stomach and then your lungs with air while breathing in; (B) Feel the expansion in the stomach; (C) Make sure the muscles from your stomach to your knee are relaxed, as if you are urinating while breathing out; (D) When there is pain, perform deep abdominal breathing exercises, and take a deep breath in and hold as much as you can; (E) Try to push the baby downward; (F) You can do it by holding your breath or breathing out quite slowly from your mouth; (G) The most important point in this stage is that you should not fill up the stomach with air, and you should push downward to deliver the baby; (H) You should continue the pushing until the pain is relieved
  Arms: Intervention Group

SUMMARY:
To determine effectiveness of breathing exercises for pregnant women during the second stage of labor on maternal pain, duration of labor, dyspnea, oxygen saturation (SPO2) and the first-minute Appearance, Pulse, Grimace, Activity and Respiration (APGAR) scores

DETAILED DESCRIPTION:
This study is about to determine effectiveness of breathing exercises for pregnant women during the second stage of labor on maternal pain, duration of labor, dyspnea, oxygen saturation SPO2 and the first-minute Appearance, Pulse, Grimace, Activity and Respiration (APGAR) scores.

Two sessions will be given to pregnant women in Intervention group. One session breathing exercises training will be given during first stage of labor by the investigator. During training all participants in Intervention group will be instructed to perform breathing exercises during the second stage of labor. The main components of breathing exercises during training will be as fellows (A) First, fill your stomach and then your lungs with air while breathing in; (B) Feel the expansion in the stomach; (C) Make sure the muscles from your stomach to your knee are relaxed, as if you are urinating while breathing out; (D) When there is pain, perform deep abdominal breathing exercises, and take a deep breath in and hold as much as you can; (E) Try to push the baby downward; (F) You can do it by holding your breath or breathing out quite slowly from your mouth; (G) The most important point in this stage is that you should not fill up the stomach with air, and you should push downward to deliver the baby; (H) You should continue the pushing until the pain is relieved. The participants will be observed during second stage of labor and their breathing will be monitored.

1. During the second stage of labor maternal labor pain will be assessed by Visual Analogue Scale.
2. Duration of second stage of labor will be counted by turning on the stop watch on the start of second stage and it will be stopped at the end when baby will be delivered.
3. Dyspnea will be monitored by dyspnea scale after performing breathing exercises during second stage of labor.
4. Oxygen saturation will be monitored by pulse oximeter during second stage of labor.
5. APGAR score of newborn will be marked in 1st minute after the birth.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females
* Gestational age ranging between 37 and 42 weeks

Exclusion Criteria:

Women using analgesics or anesthetics, Women with clinical instability Women with psychiatric disorders

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 264 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog scale | 1 day (First Visit)
  Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.
Stop watch | 1 day (First Visit)
  A stopwatch is a handheld timepiece designed to measure the amount of time that elapses between its activation and deactivation.
DYSPNEA SCALE | 1 day (First Visit)
  Dyspnea Scale quantifies disability attributable to breathlessness, and is useful for characterizing baseline dyspnea in patients with respiratory diseases.
PULSE OXIMETER | 1 day (First Visit)
  Pulse oximeter is a noninvasive instrument for monitoring a person's oxygen saturation.
APGAR | 1 day (First Visit)
  Apgar stands for "Appearance, Pulse, Grimace, Activity, and Respiration." In the test, five things are used to check a baby's health. Each is scored on a scale of 0 to 2, with 2 being the best score

CONTACTS AND LOCATIONS:
Overall Officials: Anam Aftab, Phd*, Principal Investigator — Riphah college of rehabilitation and allied health sciences - Rawalpindi
Locations (1):
- District headquarter hospital, Mirpur, Kashmir, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cicek S, Basar F. The effects of breathing techniques training on the duration of labor and anxiety levels of pregnant women. Complement Ther Clin Pract. 2017 Nov;29:213-219. doi: 10.1016/j.ctcp.2017.10.006. Epub 2017 Oct 18. PMID 29122264
- [Background] Amiri P, Mirghafourvand M, Esmaeilpour K, Kamalifard M, Ivanbagha R. The effect of distraction techniques on pain and stress during labor: a randomized controlled clinical trial. BMC Pregnancy Childbirth. 2019 Dec 30;19(1):534. doi: 10.1186/s12884-019-2683-y. PMID 31888543
- [Background] Davim RM, Torres Gde V, Melo ES. Non-pharmacological strategies on pain relief during labor: pre-testing of an instrument. Rev Lat Am Enfermagem. 2007 Nov-Dec;15(6):1150-6. doi: 10.1590/s0104-11692007000600015. PMID 18235958
- [Background] Lindholm A, Hildingsson I. Women's preferences and received pain relief in childbirth - A prospective longitudinal study in a northern region of Sweden. Sex Reprod Healthc. 2015 Jun;6(2):74-81. doi: 10.1016/j.srhc.2014.10.001. Epub 2014 Oct 12. PMID 25998874
- [Background] Marshall NE, Fu R, Guise JM. Impact of multiple cesarean deliveries on maternal morbidity: a systematic review. Am J Obstet Gynecol. 2011 Sep;205(3):262.e1-8. doi: 10.1016/j.ajog.2011.06.035. Epub 2011 Jun 15. PMID 22071057
- [Background] Akarsu RH, Mucuk S. Turkish women's opinions about cesarean delivery. Pak J Med Sci. 2014 Nov-Dec;30(6):1308-13. doi: 10.12669/pjms.306.5748. PMID 25674129
- [Background] Gonen R, Tamir A, Degani S. Obstetricians' opinions regarding patient choice in cesarean delivery. Obstet Gynecol. 2002 Apr;99(4):577-80. doi: 10.1016/s0029-7844(01)01766-5. PMID 12039114
- [Background] Lowe NK. The nature of labor pain. Am J Obstet Gynecol. 2002 May;186(5 Suppl Nature):S16-24. doi: 10.1067/mob.2002.121427. PMID 12011870
- [Background] Boaviagem A, Melo Junior E, Lubambo L, Sousa P, Aragao C, Albuquerque S, Lemos A. The effectiveness of breathing patterns to control maternal anxiety during the first period of labor: A randomized controlled clinical trial. Complement Ther Clin Pract. 2017 Feb;26:30-35. doi: 10.1016/j.ctcp.2016.11.004. Epub 2016 Nov 11. PMID 28107846
- [Background] Yildirim G, Sahin NH. The effect of breathing and skin stimulation techniques on labour pain perception of Turkish women. Pain Res Manag. 2004 Winter;9(4):183-7. doi: 10.1155/2004/686913. PMID 15605131
- [Background] Tranquilli AL, Biagini A, Greco P, Di Tommaso M, Giannubilo SR. The correlation between fetal bradycardia area in the second stage of labor and acidemia at birth. J Matern Fetal Neonatal Med. 2013 Sep;26(14):1425-9. doi: 10.3109/14767058.2013.784263. Epub 2013 Apr 17. PMID 23488805
- [Background] Schiano MA, Hauth JC, Gilstrap LC 3rd. Second-stage fetal tachycardia and neonatal infection. Am J Obstet Gynecol. 1984 Mar 15;148(6):779-81. doi: 10.1016/0002-9378(84)90566-0. PMID 6702948
- [Background] McNamara H, Johnson N. The effect of uterine contractions on fetal oxygen saturation. Br J Obstet Gynaecol. 1995 Aug;102(8):644-7. doi: 10.1111/j.1471-0528.1995.tb11403.x. PMID 7654643
- [Background] Edelstone DI, Peticca BB, Goldblum LJ. Effects of maternal oxygen administration on fetal oxygenation during reductions in umbilical blood flow in fetal lambs. Am J Obstet Gynecol. 1985 Jun 1;152(3):351-8. doi: 10.1016/s0002-9378(85)80226-x. PMID 4003479
- [Background] Davim RM, Torres Gde V, Dantas Jda C. [Effectiveness of non-pharmacological strategies in relieving labor pain]. Rev Esc Enferm USP. 2009 Jun;43(2):438-45. doi: 10.1590/s0080-62342009000200025. Portuguese. PMID 19655687
- [Background] Milne JA, Howie AD, Pack AI. Dyspnoea during normal pregnancy. Br J Obstet Gynaecol. 1978 Apr;85(4):260-3. doi: 10.1111/j.1471-0528.1978.tb10497.x. PMID 638094
- [Background] Bernardi L, Spadacini G, Bellwon J, Hajric R, Roskamm H, Frey AW. Effect of breathing rate on oxygen saturation and exercise performance in chronic heart failure. Lancet. 1998 May 2;351(9112):1308-11. doi: 10.1016/S0140-6736(97)10341-5. PMID 9643792